CLINICAL TRIAL: NCT00371813
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Multinational Study Of Efficacy And Safety Of Varenicline Tartrate For Smoking Cessation
Brief Title: An Investigation of Effectiveness and Safety of Varenicline Tartrate in Helping People Quit Smoking
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051055
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: Varenicline tartrate
Drug: Placebo

SUMMARY:
To investigate safety and efficacy of varenicline tartrate in helping people quit smoking

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smokers between the ages of 18 and 75 years, who are motivated to stop smoking

Exclusion Criteria:

* Patients currently suffering from depression, or have been diagnosed with depression in the last 12 months, or subjects with past or present history of psychosis, panic disorder, or bipolar disorder
* Any subject with known severe chronic obstructive pulmonary disease (COPD)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2006-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To compare 12 weeks of treatment with varenicline 1 mg BID to placebo for smoking cessation, and to evaluate continuous abstinence from smoking for 12 weeks after the treatment period.

SECONDARY OUTCOMES:
To gather safety data for 12 weeks of treatment with varenicline 1 mg BID or placebo followed by 12 weeks of non-treatment follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- China (6):
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Guangzhou
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Shenyang
  - Pfizer Investigational Site, Tanjin
- Pfizer Investigational Site, Singapore, Singapore
- Thailand (2):
  - Pfizer Investigational Site, Bangkok
  - Pfizer Investigational Site, Chiang Mai

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Wang C, Xiao D, Chan KP, Pothirat C, Garza D, Davies S. Varenicline for smoking cessation: a placebo-controlled, randomized study. Respirology. 2009 Apr;14(3):384-92. doi: 10.1111/j.1440-1843.2008.01476.x. Epub 2009 Feb 20. PMID 19192221
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051055&StudyName=An%20investigation%20of%20effectiveness%20and%20safety%20of%20varenicline%20tartrate%20in%20helping%20people%20quit%20smoking